CLINICAL TRIAL: NCT03967119
Title: Assessments of Dynamic Variables of Fluid Responsiveness to Predict Desufflation-induced Hypotension in Urologic Patients Undergoing Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0203
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Deflation Induced Hypotension; Laparoscopic Surgery
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic surgery: The following parameters are assessed and recorded at the following time points in all participants.
  The parameters assessed: mean arterial pressure, heart rate, pulse oxygen saturation, SVV, PPV, PWV, peak inspiratory pressure, plateau pressure, positive end-expiratory pressure, respiratory rate (all dynamic variables are assessed at two levels of tidal volume- 6 ml/kg and 12 ml/kg).
  The time points: T0, before anesthetic induction; T1, immediately after anesthetic induction; T2, immediately after pneumoperitoneum; T3, 10 min before desufflation; T4, immediately after desufflation.
  The desufflation-induced hypotension is defined as more than 20 % decrease in MAP at T4 from MAP at T3.
  Interventions: Device: Patient monitoring

INTERVENTIONS:
Device: Patient monitoring — Arterial blood pressure, pulse oxygen saturation, and cardiac output/stroke volume are monitored with invasive arterial catheter, pulse oxymetry, and esophageal doppler in all participants. Some dynamic variables including SVV and PPV are automatically calculated in each monitor. PWV is manually calculated in a printed plethysmographic waveform. Plethysmographic waveform amplitude (PW) is measured on a beat-to-beat basis as the vertical distance between peaks and preceding valley troughs in the waveform. The maximum PW (PWmax) and minimum PW (PWmin) are determined manually over the same respiratory cycle, and PWV is calculated. PWV=(PWmax-PWmin)/[(PWmax+PWmin)/2].

SUMMARY:
Laparoscopic surgery can induce hemodynamic pertubations. Pneumoperitoneum, inevitable in laparoscopic surgery, induces increase in intra-abdominal pressure, which can decrease cardiac output. Simultaneously, pneumoperitoneum can stimulate sympathetic system and increase vascular resistance/arterial blood pressure. Patients undergoing laparoscopic surgery may show a normal range of blood pressure during pneumoperitoneum even when the patients are in hypovolemia, and desufflation at the end of main surgical procedure can cause an abrupt hypotension revealing hypovolemia. Therefore, appropriate fluid management is essential for preventing desufflation-induced hypotension in laparoscopic surgery. Recently, dynamic variables are used to predict and guide fluid therapy during controlled ventilation. these variables arise from heart-lung interactions during positive ventilation, which influence left ventricular stroke volume. Several dynamic variables are derived from variations in left ventricular stroke volume (stroke volume variation, SVV), for example pulse pressure variation (PPV), and variations in pulse oximetry plethysmography waveform amplitude (PWV), which have all been shown to predict fluid responsiveness in different clinical and experimental settings. However, there are few evidences regarding which type of dynamic variables can predict desufflation-induced hypotension in laparoscopic surgery. Therefore, this study was designed to assess the predictive abilities of three different type of dynamic variables including PPV, SVV, and PWV for desufflation-induced hypotension in patients undergoing laparoscopic surgery.

DETAILED DESCRIPTION:
The study is a prospective, single-arm, and observational one. Eighty Patients who age more than 19 years and are undergoing laparoscopic surgery for urologic procedures are being enrolled in this study. All anesthetic and surgical managements are being performed according to the institutional standards. An attending anesthesiologist who is independent from this study performs anesthetic managements for the participants including fluid administration.

Investigators assess and record the following parameters at the following time points.

The parameters assessed: mean arterial pressure, heart rate, pulse oxygen saturation, SVV, PPV, PWV, peak inspiratory pressure, plateau pressure, positive end-expiratory pressure, respiratory rate (all dynamic variables are assessed at two levels of tidal volume- 6 ml/kg and 12 ml/kg).

The time points: T0, before anesthetic induction; T1, immediately after anesthetic induction; T2, immediately after pneumoperitoneum; T3, 10 min before desufflation; T4, immediately after desufflation.

The desufflation-induced hypotension is defined as more than 20 % decrease in MAP at T4 from MAP at T3.

ELIGIBILITY:
Inclusion Criteria:

* 1. laparoscopic nephrectomy
* 2. laparoscopic nephro-ureterectomy
* 3. laparoscopic adrenalectomy

Exclusion Criteria:

* 1. ASA physical status 3 and greater
* 2. preoperative arrhythmia
* 3. moderate to severe valvular disease
* 4. ventricular ejection fraction < 40%
* 5. inotrope use
* 6. moderate to severe chronic obstructive pulmonary disease
* 7. moderate to severe renal or hepatic disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic surgery for urologic procedures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
AUC for dynamic variables to predict deflation-induced hypotension | Dynamic variables at T3 (10 minutes before desufflation)
  To test the abilities of dynamic variables to predict curves (AUC) are calculated in each type of dynamic variables at each tidal volume level (6 or 12 ml/kg).
AUC for dynamic variables to predict deflation-induced hypotension | Hypotension occurence at T4 (immediately after desufflation)
  To test the abilities of dynamic variables to predict desufflation-induced hypotension, the areas under receiver-operating characteristic curves (AUC) are calculated in each type of dynamic variables at each tidal volume level (6 or 12 ml/kg).

SECONDARY OUTCOMES:
Cut-off value for dynamic variables to predict deflation-induced hypotension | Dynamic variables at T3 (10 minutes before desufflation)
  To apply dynamic variables to predict desufflation-induced hypotension into clinical practice, the cut-off values are calculated in each type of dynamic variables at each tidal volume level (6 or 12 ml/kg).
Cut-off value for dynamic variables to predict deflation-induced hypotension | Hypotension occurence at T4 (immediately after desufflation)
  To apply dynamic variables to predict desufflation-induced hypotension into clinical practice, the cut-off values are calculated in each type of dynamic variables at each tidal volume level (6 or 12 ml/kg).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei universiy college of medicine, Seoul, South Korea